CLINICAL TRIAL: NCT01014234
Title: Rapamycin and Regulatory T Cells in Renal Transplant Patients: a Two-year Randomized Prospective Study
Brief Title: Rapamycin and Regulatory T Cells in Kidney Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Carmelo Libetta, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20070034809
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Kidney Transplantation
Keywords: Immunosuppressive Agents; Immune system regulation; Regulatory T cells; Rapamycin; Tolerance
MeSH Terms: interventions — Cyclosporins; Cyclosporine; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rapamycin (Experimental): Maintenance treatment with rapamycin + mycophenolate + prednisone. This treatment will be introduced one month after renal transplantation.
  Interventions: Drug: Rapamycin
- cyclosporine (Active Comparator): Maintenance treatment with cyclosporine + mycophenolate + prednisone. This treatment will be introduced one month after renal transplantation.
  Interventions: Drug: Cyclosporins

INTERVENTIONS:
Drug: Cyclosporins — These patients will undergo maintenance immunosuppressive treatment with cyclosporine + mycophenolate + prednisone according to established clinical practice. The dosage of drugs will be based on evaluations of serum trough levels and it will be adjusted when necessary.
  Other Names: Neoral
  Arms: cyclosporine
Drug: Rapamycin — These patients will undergo maintenance immunosuppressive treatment with rapamycin + mycophenolate + prednisone according to established clinical practice. The dosage of drugs will be based on evaluations of serum trough levels and it will be adjusted when necessary.
  Other Names: Sirolimus; Rapamune
  Arms: Rapamycin

SUMMARY:
The immune system response is mediated by the interaction between the antigen presenting cell (APC), CD4+ T helper cells (Th) and CD4+ CD25+ regulatory T cells, a subgroup of CD4+ T cell which express IL-2 receptor (CD25) and the transcriptional factor foxp3. Regulatory T cell may contribute to the maintenance of tolerance by suppressing the immune response to normal or tumor associated antigens.

Regulatory T cell emerge from the thymus during ontogenesis and they represent about 10 % of the peripheral Cd4+ t cells.

Rapamycin is one the most use treatment to prevent renal allograft failure. Differently from calcineurin inhibitors (cyclosporine and tacrolimus), that inhibit T-cell activation through the inhibition of calcineurin activation, rapamycin inhibits cellular proliferation by impairing the progression of the cellular cycle, in particular by interaction with mTOR. Recently Battaglia et al. have demonstrated a Treg amplification in murine CD4+ lymphocytes treated with rapamycin in vitro.

Aim of the study is to evaluate the effect of different immunosuppressive regimens on regulatory T cell and to verify the hypothesis that rapamycin may induce tolerance in kidney transplanted patients, more than cyclosporine treatment.

DETAILED DESCRIPTION:
It is two years randomised controlled trial in parallel groups.

It has been resolved to compare different immunosuppressive regimens:

1. cyclosporine+ mycophenolate+prednisone
2. rapamycin + mycophenolate + prednisone, this treatment should be introduced after one month from renal transplantation.

Patient should visited at month 1-6-12-24 from the transplant. During the control we will reported the following data: physical examination, blood test (blood count, creatinin, BUN, immunosuppressive blood concentration, histological response of surveillance renal biopsy), blood pressure, attendant change of current therapy, pathological variation, or any hospitalisation both ordinary or in DH regimen.

Moreover in all control visit it will be collected a blood sample for evaluation of regulatory t cells.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged from 18 to 75 years
* Transplanted patients from cadaveric donors
* Patients who has given written informed consensus

Exclusion Criteria:

* Legally unable patients
* Patients who have been participated to others studies in the last 3 months
* Addicted to alcohol or smoking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The absolute number of T-reg after renal transplant in patients in treatment with rapamycin compared to patients treated with cyclosporine | Every 6 months after the transplantation

SECONDARY OUTCOMES:
Adverse events developed during the duration of the clinical study, that damage the patient, that is not part of the natural history of the disease. | Every two months during the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Dal Canton, MD, Principal Investigator — Policlinico Fondazione IRCCS "San Matteo", Pavia
Locations (1):
- Policlinico Fondazione IRCCS "San Matteo", Pavia, Italy

REFERENCES:
- [Background] Battaglia M, Stabilini A, Migliavacca B, Horejs-Hoeck J, Kaupper T, Roncarolo MG. Rapamycin promotes expansion of functional CD4+CD25+FOXP3+ regulatory T cells of both healthy subjects and type 1 diabetic patients. J Immunol. 2006 Dec 15;177(12):8338-47. doi: 10.4049/jimmunol.177.12.8338. PMID 17142730
- [Background] San Segundo D, Fernandez-Fresnedo G, Ruiz JC, Rodrigo E, Benito MJ, Arias M, Lopez-Hoyos M. Two-year follow-up of a prospective study of circulating regulatory T cells in renal transplant patients. Clin Transplant. 2010 May-Jun;24(3):386-93. doi: 10.1111/j.1399-0012.2009.01086.x. Epub 2009 Sep 11. PMID 19744094
- [Background] Ramirez E, Morales JM, Lora D, Mellado M, Cevey M, Alfaro FJ, De Pablos P, Andres A, Paz-Artal E, Serrano A. Peripheral blood regulatory T cells in long-term kidney transplant recipients. Transplant Proc. 2009 Jul-Aug;41(6):2360-2. doi: 10.1016/j.transproceed.2009.05.007. PMID 19715919